CLINICAL TRIAL: NCT02049827
Title: Evaluation of a Predictive Immunovirological Test Occurrence of BK Virus Nephropathy in Renal Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-AOI-03
Record Dates: First submitted 2014-01-28; First posted 2014-01-30 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Renal Transplant
Keywords: Renal transplant, BK virus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Renal transplant (Experimental)
  Interventions: Other: participation in the study

INTERVENTIONS:
Other: participation in the study

SUMMARY:
Kidney transplantation is the treatment of choice for end stage renal disease (ESRD) improving the quantity and quality of life for dialysis patients. Although prolongation of graft survival in the short term by preventing the release is observed by immunosuppression (IS) powerful, the longer-term survival has not improved . Indeed, the IS can not only have a direct deleterious effect on the kidney transplant , but too weak IS can promote rejection, and too strong, promote the emergence of a viral disease polyomavirus BK ( BKV ) . BK nephropathy (BKVAN ) virus is accompanied by an irreversible impairment of the renal function , leading to a loss of the graft followed by a premature return to dialysis in at least 50 % of cases. Plasma BKV reactivation was observed mainly during the first year of transplantation in 15% of patients and complications annually BKVAN concern about 5 % of recipients . Currently , treatment options are very limited , only the decrease in IS shows a partially effective when care is early . There is no specific antiviral effective treatment of this disease . In addition, there is no way to predict which patients will develop BKV reactivation BKVAN despite lower tax.

The diagnosis of interstitial nephritis BKV based on the detection of viral DNA by PCR and plasma is confirmed by histological analysis of renal tissue . Plasma quantitative PCR ( qPCR) to measure the progression of the disease and therapeutic efficacy. Control of BKV viremia is the direct antiviral immune response quality based primarily on a very effective anti- T lymphocyte activity BKV reflection. In this context, the inhibition of lymphocyte activation induced by IS blocks the establishment of T-cell responses anti- BKV in most transplant, a very low presence of T lymphocytes is generally observed in these patients anti- BKV (LYT - BKV) blood .

Our preliminary studies have validated in vitro a sensitive test to measure the functionality of blood LYT - BKV. This test is used to evaluate the concentration and functionality of LYT - BKV present in small volume of blood by measuring their specific proliferation after stimulation with peptide cocktails BKV. Proof of concept of the feasibility of this test was established on a small series of samples and highlights significant differences in lymphocyte anti-BKV different patients.

Put to good use during the post-transplant follow-up, this type of test can provide the clinician with valuable data to assess the quality of anti- BKV T response compared to the intensity and type of IS treatment. Early identification of patients at risk of reactivation of BKV, or at risk of BKVAN if BKV viremia observed , would adapt the therapeutic response and monitoring arrangements at the fair. The objective of this project is to conduct a feasibility study to assess the relevance of post-transplant monitoring of anti- BKV T response of BKV viremic patients during the first year post- transplant. Immunological data will be analyzed in relation to virological data and bioclinical data.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant > 12 months
* positive for BKV viremia
* immunosuppressive therapy including tacrolimus and mycophenolate

Exclusion Criteria:

* immunosuppressive therapy including cyclosporine and / or mTOR inhibitor
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-02-19 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Measure of BKV viral | at 6 months and 12 months
  Quantitative Measurement of BKV viral load decline after IS. Negativation sign healing, persistence is poor prognosis.

SECONDARY OUTCOMES:
stability, decrease, increase of viremia | 4 weeks, 8 weeks, 12 weeks, 6 months and 1 year
  The evolution of viremia (stability, decrease, increase) profile may also be considered to analyze the immunological data obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Laetitia ALBANO, MD, Study Director — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France